CLINICAL TRIAL: NCT06485700
Title: Peers and Technology for Adherence, Access, Accountability, and Analytics (PT4A)
Acronym: PT4A
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 24-00277
Record Dates: First submitted 2024-06-27; First posted 2024-07-03 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Cardiovascular Disease; Hypertension
MeSH Terms: conditions — Cardiovascular Diseases; Hypertension

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PT4A (Experimental): Peer delivery of medications supported by Health Information Technology (HIT) platform.
  Interventions: Other: Peer Delivery of Medications; Other: Health Information Technology (HIT) Platform
- Control (No Intervention): Participants in the control arm will receive the standard of care for hypertension or the standard of care including peer-delivery of medication.

INTERVENTIONS:
Other: Peer Delivery of Medications — Door-to-door peer delivery of medications within patients' communities will be implemented.
  Arms: PT4A
Other: Health Information Technology (HIT) Platform — The HIT platform provides: 1) tailored counseling strategies through decision support; 2) teleconsultation support for clinician-peer-patient interactions; 3) medication refill tracking to enhance accountability of the peer delivery process; and 4) analytics to improve medication supply chain by generating patient-level drug consumption data.
  Arms: PT4A

SUMMARY:
Peer-based medication delivery decreases the cost of transportation and the opportunity cost of travel while HIT can support peer activities by facilitating targeted adherence counseling, teleconsultation, synchronization of clinical care, and pharmacy activities. The investigators have implemented a pilot program of door-to-door peer-based medication delivery and HIT in western Kenya, and preliminary data indicate improved adherence and blood pressure. However, the effectiveness of this implementation strategy is not fully established. Therefore, the objective of the study is to use the PRECEDE-PROCEED framework to conduct transdisciplinary implementation research to test the hypothesis that integrating peer delivery of medications with HIT (PT4A) improves medication adherence and reduces blood pressure among patients with uncontrolled hypertension in western Kenya.

DETAILED DESCRIPTION:
Aim 1 will evaluate the effectiveness of PT4A by conducting a two-arm cluster randomized controlled implementation research hybrid type 2 trial, comparing PT4A to control. The primary biological outcome is one-year change in systolic blood pressure. The primary adherence outcome is the pill count adherence ratio. The primary implementation outcome is fidelity. Secondary outcomes are blood pressure control, self-reported adherence, and RE-AIM metrics. Aim 2 will evaluate potential mechanistic relationships between implementation measures and outcomes. Sub Aim 2.1 will evaluate if trust in the health system and patient activation mediate the relationship between PT4A and the outcomes. Aim 3 will consist of cost-effectiveness, budget impact, and qualitative analyses to help inform adaptation of PT4A to other settings. The research will be conducted by a transdisciplinary team with diverse and complementary expertise. The investigators intend to add to existing knowledge of innovative and scalable strategies to improve medication adherence for global hypertension control.

ELIGIBILITY:
Inclusion Criteria:

• Adult participants enrolled in AMPATH's CDM Program with uncontrolled hypertension (SBP ≥ 140 or diastolic BP (DBP) ≥ 90)

Exclusion Criteria:

* hypertensive emergency requiring immediate medical attention,
* terminal illness, and
* inability to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1140 (Estimated)
Dates: Start 2025-04-30 (Estimated); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Mean Change in SBP from Baseline to Month 12 | Baseline, Month 12
Pill Count Adherence Ratio (PCAR) at Month 12 | Month 12
  PCAR is calculated as the percentage of pills taken over the previous month and is measured over a 30-day time period.
Number of Patient E-Signatures | Up to Month 12
  Measure of fidelity.
Number of Completed HIT Forms | Up to Month 12
  Measure of fidelity.

SECONDARY OUTCOMES:
Mean Change in SBP from Baseline to Month 6 | Baseline, Month 6
Percentage of Participants with Controlled Blood Pressure (BP) at Month 6 | Month 6
  BP measured using automatic BP monitor.
Percentage of Participants with Controlled BP at Month 12 | Month 12
  BP measured using automatic BP monitor.

CONTACTS AND LOCATIONS:
Overall Officials: Rajesh Vedanthan, Principal Investigator — NYU Langone Health
Locations (3):
- Kenya (3):
  - Study Site, Webuye, Bungoma County
  - Study Site, Kitale, Trans Nzoia County
  - Study Site, Eldoret, Uasin Gishu County

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to: Rajesh.vedanthan@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research
Access Criteria: The investigator who proposed to use the data will be granted access upon reasonable request. Requests should be directed to Rajesh.vedanthan@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.